CLINICAL TRIAL: NCT02432300
Title: The Emotion Builder: An Intervention for Emotional Deficits After Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EmotEd (Industry)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Dawn Neumann, Assistant Research Professor, Department of Physical Medicine and Rehabilitation, IU School of Medicine, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R41HD077967-01A1 (NIH); 1404681990 (Other: Institutional Review Board (IRB)); 1R41HD077967-01A1 (NIH)
Record Dates: First submitted 2015-04-24; First posted 2015-05-04 (Estimated); Results first posted 2017-11-22 (Actual); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Traumatic Brain Injury; Alexithymia
Keywords: Traumatic Brain Injury; Alexithymia; Emotions
MeSH Terms: conditions — Brain Injuries, Traumatic; Affective Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): Treatment sessions with a virtual treatment program called Emotion Builder
  Interventions: Behavioral: Emotion Builder

INTERVENTIONS:
Behavioral: Emotion Builder — Total of 8 therapy sessions with the Emotion Builder over approximately four (4) weeks (2 sessions a week)

SUMMARY:
The purpose of this study is to examine a web-based training program for treating emotional problems in people who have suffered a traumatic brain injury (TBI).

DETAILED DESCRIPTION:
This is a pilot study to examine how subjects with TBI feel about the virtual reality program as a treatment and to assess the effectiveness of the virtual reality program at increasing subjects' awareness and understanding of emotions.

ELIGIBILITY:
Inclusion Criteria:

* TBI (injury due to an external physical force);
* Moderate to severe TBI, defined either by74 Glasgow Coma Score at time of injury (≤12), or post-traumatic amnesia (≥1 day), or loss of consciousness (≥30 minutes);
* ≥1 year post-injury;
* between 18-65 years old;
* Have a moderate to high alexithymia score (≥52) on the TAS-2070 at screening.

Exclusion criteria:

* Diagnosed with pre-morbid neurological disorders (e.g. stroke, autism, alzheimer's disease, Parkinson's disease);
* Formerly diagnosed with a developmental disability;
* Pre-morbid diagnosis of major psychiatric disorders (e.g. schizophrenia);
* Unable to follow directions;
* Uncorrected visual or hearing impairments that would prevent sufficient task participation;
* No access to reliable transportation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-05; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Neumann, PhD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Health Facilities, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Neumann D, Malec JF, Hammond FM. Reductions in Alexithymia and Emotion Dysregulation After Training Emotional Self-Awareness Following Traumatic Brain Injury: A Phase I Trial. J Head Trauma Rehabil. 2017 Sep/Oct;32(5):286-295. doi: 10.1097/HTR.0000000000000277. PMID 28060205

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were only enrolled in the treatment if they were found to have met the criteria for moderate to severe alexithymia on the Toronto Alexithymia Scale 20 (>=52).
Groups:
- Treatment Group (Emotion Builder): The intervention was a web-based treatment program called the Emotion Builder that was delivered by a clinician research assistant individually to participants.
  Emotion Builder: Total of 8 therapy sessions (60-90 minutes each) over approximately four (4) weeks (2 sessions a week). The objective of these sessions were to increase emotional awareness and labeling. Lessons included exercises designed to build emotional vocabulary, lessons to help differentiate emotions, activities to enhance attention to changes in body states associated with emotional responses (emotional arousal), and virtual videos simulating emotional scenarios for practicing lessons learned.
Period: Overall Study
Arm/Group | Treatment Group (Emotion Builder)
Started | 17
Completed | 13
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Group (Emotion Builder)
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.12 (11.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Toronto Alexithymia Scale [Mean (Standard Deviation); unit: units on a scale] — Measures emotional awareness (difficulty identifying feelings), difficulty describing feelings, and externally oriented thinking. The full scale range is 20-100 (higher scores indicate higher alexithymia). Subscales are summed to compute a total score Scores between 52 and 60 indicate moderate alexithymia; scores 61 and higher indicate high alexithymia. Population: Because 4 participants withdrew, we provide only baseline data here for those who completed the intervention (n=13).
  units on a scale
    number analyzed (Participants) | 13
    (all) | 61.54 (7.26)
Levels of Emotional Awareness Scale [Mean (Standard Deviation); unit: units on a scale] — Participants must respond how they think they would feel and how another person would feel in response to a hypothetical scenario. The more discrete emotions (e.g., bad vs sad) receive higher points, as well as blended emotions (e.g. sad and angry). There are 10 items on this measure. The minimum score for each item is 0 and the max score for each item is 5. The item scores are summed to calculate a total score. Thus, the total scores range from 0-50; 0=lowest awareness and 50=highest awareness. A computerized scoring system and parallel forms were used. Population: Because 4 participants withdrew, we provide only baseline data here for those who completed the intervention (n=13).
  units on a scale
    number analyzed (Participants) | 13
    (all) | 36.92 (7.88)
PHQ 9 (Depression) [Mean (Standard Deviation); unit: units on a scale] — The PHQ-9 is a subjective measure of depression. There are 9 items describing problems associated with depression, and participants must rate how often they have been bothered by the problems in the last 2 weeks on a 0-3 scale. The scores are summed for a total depression score, ranging from 0-27, which higher scores indicating greater depression. Population: Because 4 participants withdrew, we provide only baseline data here for those who completed the intervention (n=13).
  units on a scale
    number analyzed (Participants) | 13
    (all) | 10.77 (4.82)
Trait Anxiety (State Trait Anxiety Inventory) [Mean (Standard Deviation); unit: T score] — The STAI is a self-report measure of state and trait anxiety (20 items each). The trait anxiety subscale was the variable of interest for this study. Higher scores indicate more trait or state anxiety. Scores for each scale range from 20-80 (higher scores indicated higher anxiety). The raw scores were converted into T scores using age and gender norms provided by the STAI authors. A T score of 50 represents the mean. A difference of 10 from the mean indicates a difference of 1 standard deviation. Higher T scores still indicated higher anxiety. We reported T scores for trait anxiety. Population: Because 4 participants withdrew, we provide only baseline data here for those who completed the intervention (n=13).
  T score
    number analyzed (Participants) | 13
    (all) | 68.38 (11.45)

OUTCOME MEASURES:

1. Primary Outcome: Toronto Alexithymia Scale-20 (TAS-20)
Description: This is a 20-item self-report questionnaire comprised of three sub-constructs (Difficulty Identifying feelings, Difficulty Describing Feelings, Externally-oriented Thinking). The full scale range is 20-100 (higher scores indicate higher alexithymia). Subscales are summed to compute a total score Scores between 52 and 60 indicate moderate alexithymia; scores 61 and higher indicate high alexithymia.
Time Frame: Week 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group (Emotion Builder)
Number analyzed (Participants) | 13
units on a scale | 52.54 (11.95)

2. Primary Outcome: Levels of Emotional Awareness Scale (LEAS)
Description: The LEAS is comprised of ten hypothetical scenarios that are three or four sentences in length. Participants must respond how they think they would feel and how another person would feel in response to the hypothetical scenario. The more discrete emotions (e.g., bad vs sad) receive higher points, as well as blended emotions (e.g. sad and angry). There are 10 items on this measure. The minimum score for each item is 0 and the max score for each item is 5. The item scores are summed to calculate a total score. Thus, the total scores range from 0-50; 0=lowest awareness and 50=highest awareness. A computerized scoring system and parallel forms were used.
Time Frame: Week 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group (Emotion Builder)
Number analyzed (Participants) | 13
units on a scale | 44.23 (5.23)

3. Secondary Outcome: Patient Health Questionnaire-9 (PHQ-9) as an Assessment of Depression
Description: The PHQ-9 is a self-report questionnaire designed to assess depression through nine questions that come directly from the DSM-IV signs and symptoms of major depression. The 9 items describe problems associated with depression, and participants must rate how often they have been bothered by the problems in the last 2 weeks on a 0-3 scale. The scores are summed for a total depression score, ranging from 0-27, which higher scores indicating greater depression.
Time Frame: Week 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group (Emotion Builder)
Number analyzed (Participants) | 13
units on a scale | 9.69 (5.25)

4. Secondary Outcome: State Trait Anxiety Inventory (STAI)
Description: The STAI is a self-report measure of state and trait anxiety (20 items each). The trait anxiety subscale was the variable of interest for this study. Higher scores indicate more trait or state anxiety. Scores for each scale range from 20-80, with higher scores indicating greater anxiety. The raw scores were converted into T scores using age and gender norms provided by the authors for the STAI. A score of 50 represents the mean. A difference of 10 from the mean indicates a difference of one standard deviation. Higher T scores were still indicative of higher anxiety. We reported T scores for trait anxiety.
Time Frame: Week 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group (Emotion Builder)
Number analyzed (Participants) | 13
units on a scale | 61.54 (12.08)

ADVERSE EVENTS:
Time Frame: One year. From the start of participant enrollment until the last day of testing.
Groups:
- Treatment Group (Emotion Builder): 8 sessions of a web-based treatment, each lasting 60-90 minutes, twice per week over 4 weeks with a clinician research assistant. This treatment aimed to improve emotional awareness and labeling.
Arm/Group | Treatment Group (Emotion Builder)
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 1/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (Emotion Builder) (N=17)
Emotional Distress (Psychiatric disorders) | 1 (1) — Participant said that he did not like the treatment or how it made him feel.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes